CLINICAL TRIAL: NCT06083688
Title: Preventing Malaria in School Children to Protect the Whole Community in Rural Blantyre District, Malawi
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-048
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Malaria,Falciparum; Anemia in Children
Keywords: IPTsc; school; chemoprevention; intermittent preventive treatment; malaria transmission
MeSH Terms: conditions — Malaria, Falciparum | interventions — Chloroquine; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Students will be randomized to three arms Arm 1: intermittent preventive treatment with dihydroartemisinin-piperaquine (IPTsc-DP); Arm 2: intermittent preventive treatment with sulfadoxine-pyrimethamine plus amodiaquine (IPTsc-SPAQ); Arm 3 the control arm. Females 13 years and older (likely post-menarche) in Arms 1 and 2 will receive chloroquine alone.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermittent Preventive Treatment with dihydroartemisinin-piperaquine (IPT-DP) (Experimental): All students are treated at each intervention. Treatment will be with DP (females less than 13 years old and all males) or chloroquine (females 13 years old or older).
  Interventions: Drug: Dihydroartemisinin-Piperaquine; Drug: Chloroquine
- Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus amodiaquine (IPT-SPAQ) (Experimental): All students are treated at each intervention. Treatment will be with SP and AQ (females less than 13 years old and all males) or chloroquine (females 13 years old or older).
  Interventions: Drug: Chloroquine; Drug: Sulfadoxine-pyrimethamine-amodiaquine
- Control (No Intervention): Students will not receive preventive treatment.

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine — Treatment will be with DP (females less than 13 years old and all males) or chloroquine alone (females 13 years old or older).
  Other Names: DP; D-Artepp; DuoCotecxin; Artekin; Eurartesim; Ridmal
  Arms: Intermittent Preventive Treatment with dihydroartemisinin-piperaquine (IPT-DP)
Drug: Chloroquine — Treatment will be with CQ alone if female and 13 years old or older in both intervention arms.
  Other Names: Aralen; Hydroxychloroquine; Lariago
  Arms: Intermittent Preventive Treatment with dihydroartemisinin-piperaquine (IPT-DP); Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus amodiaquine (IPT-SPAQ)
Drug: Sulfadoxine-pyrimethamine-amodiaquine — Treatment in Arm 2 (females less than 13 years old and all males).
  Other Names: SPAQ; SPAQ-Co
  Arms: Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus amodiaquine (IPT-SPAQ)

SUMMARY:
This is an individually randomized, controlled, single blind three arm clinical trial of malaria chemoprevention strategies Arm 1: Intermittent preventive treatment with dihydroartemisinin-piperaquine (IPT-DP). Arm 2: Intermittent preventive treatment with sulfadoxine-pyrimethamine (SP) plus amodiaquine (AQ) (IPT-SPAQ). Arm 3: Control - students will receive standard of care (no preventive treatment). Outcomes include P. falciparum infection and parasite density, anemia, cognitive function and educational testing, as well as infection prevalence and disease incidence in young children sleeping student's households to assess the impact on transmission.

DETAILED DESCRIPTION:
Students attending primary school in rural Blantyre District, Malawi will be offered enrollment in this study. The intervention will be conducted every 6-weeks during the school terms which coincide with peak malaria transmission. Students in the IPT-DP arm will be treated with with dihydroartemisinin-piperaquine (DP) (females less than 13 years old and all males) or chloroquine (females 13 years old or older). Students in the IPT-SPAQ arm will be treated with sulfadoxine-pyrimethamine plus amodiaquine (females less than 13 years old and all males) or chloroquine alone (females 13 years old or older). Students in the all arms will receive routine malaria education.

ELIGIBILITY:
Student Inclusion Criteria:

* Currently enrolled in the study school
* Plan to attend the study school for the remainder of the school year
* Parent/guardian available to provide written informed consent

Student Exclusion Criteria:

* Current evidence of severe malaria or danger signs
* Known adverse reaction to the study drugs
* History of cardiac problems or fainting
* Taking medications known to prolong QT
* Family history of prolonged QT
* History of epilepsy or psoriasis
* Taking cotrimoxazole for long-term prophylaxis

Younger child Inclusion Criteria

* Slept in the household for most nights in the last month
* Age 6-59 months
* Parent/guardian available to provide written informed consent

Younger child Exclusion Criteria

- Current evidence of severe malaria or danger signs

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with P. falciparum infection | 6-8 weeks after the last intervention
  detected by polymerase chain reaction (PCR, binary)
Number of participants with anemia | 6-8 weeks after the last intervention
  World Health Organization age-sex definitions (binary)
Rate of clinical malaria | through study completion (approximately 6 months), and 6 months following the intervention
  cumulative incidence

SECONDARY OUTCOMES:
Mean hemoglobin concentration | 6-8 weeks after the last intervention
  g/dL (continuous)
Literacy skills | 6-8 weeks after the last intervention
  Early grade reading assessment
Math skills | 6-8 weeks after the last intervention
  Early grade math assessment
Rate of school absenteeism among participants | through study completion (approximately 6 months)
  Proportion of days absent among days where attendance is assessed
P. falciparum prevalence among children less than 5 years old living in households with study participants | 6-8 weeks after the last intervention
  detected by PCR
Rate of clinical malaria among children less than 5 years old living in households with study participants | through study completion (approximately 6 months)
  cumulative incidence

OTHER OUTCOMES:
Total parasite density | 6-8 weeks after the last intervention
  log transformed (continuous)

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Alert Centre, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: After publication
Access Criteria: Public access with registration to allow tracking